CLINICAL TRIAL: NCT01294423
Title: A 24-week Randomised, Double-blind, Parallel-group, Multi-centre, Placebo-controlled Phase III Trial to Evaluate the Efficacy and Safety of Dapagliflozin as Monotherapy in Japanese Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise
Brief Title: Evaluate Efficacy and Safety in Japanese Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1692C00006
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Type 2 Diabetes; High Blood Sugar
Keywords: Phase3; Clinical trial; Type2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Dapagliflozin 5 mg
  Interventions: Drug: Dapagliflozin
- 2 (Experimental): Dapagliflozin 10 mg
  Interventions: Drug: Dapagliflozin
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 5mg/matching placebo for Dapagliflozin 10mg oral dose
  Arms: 1
Drug: Dapagliflozin — Dapagliflozin 10mg/matching placebo for Dapagliflozin 5mg oral dose
  Arms: 2
Drug: Placebo — Matching placebo for Dapagliflozin 5mg/10mg oral dose
  Arms: 3

SUMMARY:
This is a 24-week randomised, multi-centre phase III study to evaluate the efficacy and safety of dapagliflozin as monotherapy in Japanese subjects with Type 2 diabetes mellitus who have inadequate glycemic control with diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Men or women age ≥20 years old (Either gender needs to be 40% or higher of total number of treated subjects)diagnosed with type 2 DM ; ≥6.5% and ≤10% at 1 week before randomization

Exclusion Criteria:

* Type 1 diabetes mellitus
* FPG >240 mg/dL before randomization
* Subjects who have history of unstable or rapidly progressing renal disease
* Subjects who have severe hepatic insufficiency and/or significant abnormal liver function
* Significant cardiovascular history

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jisin Yang, MD, Study Director — AstraZeneca KK
Locations (26):
- Japan (26):
  - Research Site, Noda, Chiba
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Yukuhashi, Fukuoka
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Chitose-shi, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Takasago-shi, Hyōgo
  - Research Site, Hakusan-shi, Ishikawa-ken
  - Research Site, Sanuki-shi, Kagawa-ken
  - Research Site, Takamatsu, Kagawa-ken
  - Research Site, Ebina-shi, Kanagawa
  - Research Site, Kamakura-shi, Kanagawa
  - Research Site, Sendai, Miyagi
  - Research Site, Matsumoto-shi, Nagano
  - Research Site, Okayama, Okayama-ken
  - Research Site, Osaka, Osaka
  - Research Site, Suita, Osaka
  - Research Site, Ōtsu, Shiga
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Chuo-ku, Tokyo
  - Research Site, Chūō, Tokyo
  - Research Site, Meguro-ku,, Tokyo
  - Research Site, Ōta-ku, Tokyo
  - Research Site, Tokyo, Tokyo
  - Research Site, Takaoka-shi, Toyama
  - Research Site, Toyama, Toyama

REFERENCES:
- [Background] Kaku K, Kiyosue A, Inoue S, Ueda N, Tokudome T, Yang J, Langkilde AM. Efficacy and safety of dapagliflozin monotherapy in Japanese patients with type 2 diabetes inadequately controlled by diet and exercise. Diabetes Obes Metab. 2014 Nov;16(11):1102-10. doi: 10.1111/dom.12325. Epub 2014 Jul 8. PMID 24909293
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=298&filename=CSR-D1692C00006.pdf
- See also: CSR-D1692C00006.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=298&filename=CSR-D1692C00006.pdf
- See also: D1692C00006_Clinical_Study_Protocol_and_Amendment — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=298&filename=D1692C00006_Clinical_Study_Protocol_and_Amendment_8536419317510300265.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled: 25 Feb 2011. Last participant completed 24 week period: 12 Mar 2012. 354 participant were enrolled in 30 Japanese centers. 261 participants were randomized. Japanese men or women aged >= 20 years with inadequate glycemic control (HbA1c 6.5% to 10.0%) with diet and exercise.
Pre-assignment Details: Wash-out period was applicable only for participants with ongoing anti-diabetic treatment at enrolment. Drug-naive participants skip the period and directly proceed to a placebo lead-in period.
Groups:
- Dapagliflozin 5 mg: Dapagliflozin : Dapagliflozin 5mg/matching placebo for Dapagliflozin 10mg oral dose
- Dapagliflozin 10 mg: Dapagliflozin : Dapagliflozin 10mg/matching placebo for Dapagliflozin 5mg oral dose
- Placebo: Placebo : Matching placebo for Dapagliflozin 5mg/10mg oral dose
Period: Overall Study
Arm/Group | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Placebo
Started | 86 | 88 | 87
Completed | 81 | 79 | 79
Not Completed | 5 | 9 | 8
Not completed — Adverse Event | 1 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — subject no longer meets study criteria | 2 | 5 | 2
Not completed — poor/non-compliance | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Placebo | Total
Number analyzed (Participants) | 86 | 88 | 87 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.41) | 57.5 (9.29) | 60.4 (9.65) | 58.9 (9.83)
Age, Customized [Number; unit: participants]
  < 65 years | 59 | 67 | 55 | 181
  65 - <75 years | 23 | 20 | 29 | 72
  >= 75 years | 4 | 1 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 35 | 106
  Male | 50 | 53 | 52 | 155
Region of Enrollment [Number; unit: participants]
  Japan | 86 | 88 | 87 | 261
Body Weight [Mean (Standard Deviation); unit: kg] | 65.81 (14.371) | 69.70 (13.821) | 65.96 (12.908) | 67.17 (13.777)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.88 (3.907) | 26.06 (4.519) | 25.22 (4.394) | 25.39 (4.296)
Seated Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 122.0 (13.01) | 126.2 (12.46) | 126.5 (14.36) | 124.9 (13.41)
HbA1c [Mean (Standard Deviation); unit: Percent] | 7.50 (0.718) | 7.46 (0.608) | 7.50 (0.625) | 7.49 (0.649)
FPG [Mean (Standard Deviation); unit: mg/dL] | 137.5 (24.41) | 138.8 (22.14) | 139.6 (21.63) | 138.6 (22.68)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: To compare change from baseline in HbA1c achieved with each dose of dapagliflozin versus placebo after 24 weeks double-blind treatment.
Time Frame: From Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 86 | 87 | 86
Percent | -0.41 [-0.53 to -0.29] | -0.45 [-0.57 to -0.33] | -0.06 [-0.18 to 0.06]
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg vs Placebo; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0 (with alpha = 0.027 applying Dunnett's adjustment, two-sided); Test type: Superiority or Other; p < 0.0001, ANCOVA — significant at alpha=0.027 (2-sided) applying Dunnett's adjustment. A hierarchical closed testing procedure was used to control the Type I error rate across the primary and key secondary endpoints; with treatment group (all treatment groups included) and gender as effect and baseline value as covariate; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.52 to -0.18], Standard Error of Mean 0.0853
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; with treatment group (all treatment groups included) and gender as effect and baseline value as covariate; Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.56 to -0.23], Standard Error of Mean 0.0851

2. Secondary Outcome: Adjusted Mean Change in Fasting Plasma Glucose (FPG)
Description: To compare the change from baseline in fasting plasma glucose (FPG) achieved with each dose of dapagliflozin versus placebo after 24 weeks double-blind treatment.
Time Frame: From Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 86 | 87 | 86
mg/dL | -8.6 [-12.9 to -4.3] | -13.7 [-18.0 to -9.5] | 5.8 [1.6 to 10.1]
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg vs Placebo; The null hypothesis is given as H0: mean(treat) minus mean(placebo) = 0 versus HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure within treatment group; with treatment group (all treatment groups included) and stratum (HbA1c at randomization by gender) as effect and baseline value as covariate; Mean Difference (Final Values) = -14.4, 95% CI 2-sided [-20.1 to -8.7], Standard Error of Mean 2.902
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -19.5, 95% CI 2-sided [-25.2 to -13.8], Standard Error of Mean 2.892

3. Secondary Outcome: Adjusted Mean Change in Body Weight
Description: To compare the change from baseline in total body weight achieved with each dose of dapagliflozin versus placebo after 24 weeks double-blind treatment.
Time Frame: From Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Placebo
Number analyzed (Participants) | 86 | 88 | 87
kg | -2.13 [-2.65 to -1.60] | -2.22 [-2.73 to -1.71] | -0.84 [-1.36 to -0.32]
Statistical Analysis 1: Comparison: Dapagliflozin 5 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.29, 95% CI 2-sided [-1.98 to -0.59], Standard Error of Mean 0.3533
Statistical Analysis 2: Comparison: Dapagliflozin 10 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-2.08 to -0.69], Standard Error of Mean 0.3540

ADVERSE EVENTS:
Time Frame: Non-serious/serious adverse events on or after the first day and on or prior to the last day of the 24-week double-blind treatment period plus 4/30 days or up to follow-up visit if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Dapagliflozin 5 mg | Dapagliflozin 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/86 | 1/88 | 1/87
Other Adverse Events (participants affected / at risk) | 11/86 | 15/88 | 14/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 5 mg (N=86) | Dapagliflozin 10 mg (N=88) | Placebo (N=87)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
PUTAMEN HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin 5 mg (N=86) | Dapagliflozin 10 mg (N=88) | Placebo (N=87)
NASOPHARYNGITIS (Infections and infestations) | 9 | 15 | 9
HYPERTENSION (Vascular disorders) | 2 | 1 | 5

LIMITATIONS AND CAVEATS:
For participants who did not complete 24 weeks LOCF (last observation carried forward) was used. Only values prior to rescue medication were used for outcome measures except for total body weight which was evaluated regardless of rescue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.